CLINICAL TRIAL: NCT01930669
Title: Transplanted-like Heart in Critical Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Regione Lombardia (Other)
Responsible Party: Principal Investigator, Riccardo Colombo, MD, ASST Fatebenefratelli Sacco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DR#13465/22Dec2011
Record Dates: First submitted 2013-08-14; First posted 2013-08-29 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Autonomic Nervous System Dysfunction in Critically Ill
Keywords: Heart Rate Variability; Multiple Organ Dysfunction Syndrome; Critically Ill
MeSH Terms: conditions — Multiple Organ Failure; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Other): To measure the autonomic nervous system activity elicited by a gravitational sympathetic stimulus in critically ill
  Interventions: Other: Gravitational sympathetic stimulus

INTERVENTIONS:
Other: Gravitational sympathetic stimulus — Autonomic nervous system (ANS) activity is assessed by means of HRV, SAP variability and baroreflex control analysis daily from day 1 to discharge from ICU or day 28.
  Analysis is performed (i)at rest in supine position with bed at zero degrees of inclination (ii) during modified tilt (MTILT) and (iii) recovery from MTILT in supine position at zero degrees. In a subgroup of patients motor sympathetic nervous activity (MSNA) is recorded at day 1,2 and 7.
  MTILT consists in elevating head and trunk of patients at 60 degrees and lowering legs at 15 degree with a standard critical care bed. MSNA is recorded from the external peroneal nerve with microneurographic technique.

SUMMARY:
The purpose of this study is to measure the dysfunction of the autonomic nervous system in modulating the heart rate variability and baroreflex control in critically ill.

DETAILED DESCRIPTION:
Autonomic nervous system (ANS) is able to change both heart beat-to-beat interval and peripheral muscle vascular tone in response to different stimuli. Unfortunately the direct measure of the sympathetic and vagal activity appears not feasible in a clinical setting. ANS modulation is studied non-invasively by means of heart rate variability (HRV) and baroreflex sensitivity. Decreased HRV has been found in critical ill patients with multiple organ dysfunction syndrome (MODS) and sepsis, thus it has been supposed being a sign of autonomic dysfunction. Frequently, in mechanically ventilated critical ill patients the HRV does not show any oscillatory pattern, as well as it appears in the early months after heart transplantation. Under these circumstances the heart seems to lack the neuro-modulatory control by ANS and it seems to respond exclusively to the preload and afterload laws. This could have implications for outcome because autonomic dysfunction is associated with increasing severity of illness and mortality. Since the ANS modulation is a dynamic process that implies a central integration of a complex variety of afferent stimuli (from carotid sinus, cardiopulmonary receptors, pain,…) and efferences through sympathetic and vagal branches, up to the present it is unclear if in critically ill a reduced HRV at rest reflects a state of low requirement of ANS modulation or truly a failure of the ANS. To provide new insights into this important topic we study the changes of ANS modulation in response to a orthostatic sympathetic stimulus daily from the day of ICU admission until day 28, or the day of discharge from ICU if it occurs before the day 28.

Measurements. Beat-to-beat intervals are computed detecting the QRS complex on the electrocardiogram and locating the R-apex using parabolic interpolation. The maximum arterial pressure within each R-to-R interval is taken as systolic arterial pressure (SAP). Sequences of 300 values are randomly selected inside each experimental condition. The power spectrum is estimated according to a univariate parametric approach fitting the series to an autoregressive model. Autoregressive spectral density is factorized into components each of them characterized by a central frequency. A spectral component is labeled as low frequency (LF) if its central frequency is between 0.04 and 0.15 Hz, while it is classified as high frequency (HF) if its central frequency is between 0.15 and 0.4 Hz. The HF power of R-to-R series is utilized as a marker of vagal modulation directed to the heart , while the LF power of SAP series is utilized as a marker of sympathetic modulation directed to vessels. The ratio of the LF power to the HF power assessed from R-to-R series is taken as an indicator sympatho-vagal balance directed to the heart. Baroreflex control in the low frequencies is computed as the square root of the ratio of LF(RR) to LF(SAP). In the same way baroreflex control in the high frequencies is defined as the square root of the ratio of HF(RR) to HF(SAP).

The experimental condition is a sequence of three time point each lasting 10 min: (i) rest, with patient in supine position at zero degree; (ii) modified tilt; (iii) recovery, with the patient supine.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted in ICU with

* age between 18 and 75 years
* expected length of stay in ICU >24 hours
* sinus rhythm on ECG
* ectopic heart beats <5% of all heart beats
* no contraindications of any kind to head-up 60 degrees position

Exclusion Criteria:

* age <18 and >75 years
* elective postoperative patients
* non sinusal rhythm of ECG
* ectopic heart beats >5% of all heart beats
* spinal or head injury
* suspected or documented intracranial hypertension
* contraindications of any kind to head up 60 degrees position

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of autonomic nervous system dysfunction in critical ill patients | from day 1 to day 28
  failure to change significantly HRV and baroreflex variables in response to MTILT.

SECONDARY OUTCOMES:
to measure the occurrence of ANS failure in subgroups | from day 1 to day 28
  subgroups: (i) sepsis; (ii) severe sepsis/ septic shock; (iii) failure affecting >1 organ as assessed by SOFA score; (iv) death/alive at ICU discharge We calculate the hazard ratio for each subgroup. We calculate the Cox's proportional model to identify the factors predisposing occurrence of ANS dysfunction/failure.
  ANS failure definition: see secondary outcome
Length of stay in ICU and in Hospital | 8 months
  We measure length of stay in ICU and in hospital of patients without ANS dysfunction, with ANS dysfunction and with ANS failure
mortality | 8 months
  We measure mortality among subgroups of patients ((i)without ANS dysfunction, (ii)with ANS dysfunction and (iii)with ANS failure), adjusted for severity of illness assessed with Simplified Acute Physiology Score(SAPSII)
days free from mechanical ventilation | 28 days
  We measure days free from mechanical ventilation among patients without ANS dysfunction, with ANS dysfunction and with ANS failure

OTHER OUTCOMES:
to define ANS dysfunction and failure in response to MTILT | 28 days
  First, we take the HRV and baroreflex variables' changes collected at day 1 of ICU stay in the first 50 patients. We set two cut-off values: (i)below 25th and (ii) below 10th percentiles. We define ANS dysfunction the presence of at least 1 HRV variable OR 1 baroreflex variable respectively below the first cut-off value (i), otherwise we define ANS failure the presence of at least 1 HRV variable OR 1 baroreflex variable below the second cut-off value (ii).
  Second, we prospectively test these cut-off values in the remaining 100 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinando Raimondi, Director, Study Chair — Azienda Ospedaliera "L.Sacco"; Riccardo Colombo, Consultant, Principal Investigator — Azienda Ospedaliera "L.Sacco"; Stefano Guzzetti, Director, Study Director — Azienda Ospedaliera "L.Sacco"
Locations (2):
- Italy (2):
  - Azienda Ospedaliera "Luigi Sacco" - Polo Universitario - University of Milan, Milan
  - Istituto Clinico Humanitas, Rozzano

REFERENCES:
- [Background] Mazzeo AT, La Monaca E, Di Leo R, Vita G, Santamaria LB. Heart rate variability: a diagnostic and prognostic tool in anesthesia and intensive care. Acta Anaesthesiol Scand. 2011 Aug;55(7):797-811. doi: 10.1111/j.1399-6576.2011.02466.x. Epub 2011 Jun 9. PMID 21658013
- [Background] Morris JA Jr, Norris PR, Waitman LR, Ozdas A, Guillamondegui OD, Jenkins JM. Adrenal insufficiency, heart rate variability, and complex biologic systems: a study of 1,871 critically ill trauma patients. J Am Coll Surg. 2007 May;204(5):885-92; discussion 892-3. doi: 10.1016/j.jamcollsurg.2007.01.019. Epub 2007 Mar 23. PMID 17481504
- [Background] Schmidt H, Hoyer D, Wilhelm J, Soffker G, Heinroth K, Hottenrott K, Said SM, Buerke M, Muller-Werdan U, Werdan K. The alteration of autonomic function in multiple organ dysfunction syndrome. Crit Care Clin. 2008 Jan;24(1):149-63, ix. doi: 10.1016/j.ccc.2007.10.003. PMID 18241783
- [Background] Wieske L, Kiszer ER, Schultz MJ, Verhamme C, van Schaik IN, Horn J. Examination of cardiovascular and peripheral autonomic function in the ICU: a pilot study. J Neurol. 2013 Jun;260(6):1511-7. doi: 10.1007/s00415-012-6818-6. Epub 2012 Dec 30. PMID 23275003
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900
- [Background] Pagani M, Montano N, Porta A, Malliani A, Abboud FM, Birkett C, Somers VK. Relationship between spectral components of cardiovascular variabilities and direct measures of muscle sympathetic nerve activity in humans. Circulation. 1997 Mar 18;95(6):1441-8. doi: 10.1161/01.cir.95.6.1441. PMID 9118511
- [Background] Porta A, Baselli G, Rimoldi O, Malliani A, Pagani M. Assessing baroreflex gain from spontaneous variability in conscious dogs: role of causality and respiration. Am J Physiol Heart Circ Physiol. 2000 Nov;279(5):H2558-67. doi: 10.1152/ajpheart.2000.279.5.H2558. PMID 11045994
- [Background] Furlan R, Porta A, Costa F, Tank J, Baker L, Schiavi R, Robertson D, Malliani A, Mosqueda-Garcia R. Oscillatory patterns in sympathetic neural discharge and cardiovascular variables during orthostatic stimulus. Circulation. 2000 Feb 29;101(8):886-92. doi: 10.1161/01.cir.101.8.886. PMID 10694528
- [Background] Cooke WH, Hoag JB, Crossman AA, Kuusela TA, Tahvanainen KU, Eckberg DL. Human responses to upright tilt: a window on central autonomic integration. J Physiol. 1999 Jun 1;517 ( Pt 2)(Pt 2):617-28. doi: 10.1111/j.1469-7793.1999.0617t.x. PMID 10332107